CLINICAL TRIAL: NCT04457843
Title: The Mobile COPD Status Test (mCST) - Investigation of the Correlation of a Digital Measurement With Disease Relevant Endpoints in Patients With COPD
Brief Title: The Mobile COPD Status Test (mCST)
Status: Completed | Type: Observational
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Professor for pulmonary rehabilitation, Schön Klinik Berchtesgadener Land
Other Study IDs: mCST - Kaia App
Record Dates: First submitted 2020-06-04; First posted 2020-07-07 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Telehealth; disease progression; disease activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- COPD patients
  Interventions: Other: usual medical care

INTERVENTIONS:
Other: usual medical care — Prospective monitoring of clinical Outcomes and digital collected outcomes via the mobile COPD staus test app.

SUMMARY:
Up tp now, disease activity of COPD patients in their home environment has usually been recorded by questionnaires (e.g. COPD assessment test). Digital multifactorial measurements, via the "mobile COPD Status test" app, offer a new way of displaying disease activity. However, there is no independent study that has examined whether digitally collected parameters correlate with the common used measurement instruments for COPD patients (both in cross-sectional and longitudinal course).

The aim of this exploratory study is to investigate the correlation between the mobile COPD Status test (mCST App, KAIA Health) and a conventional collected clinical data set of routine measurements as well as the subjective symptoms and activity perception of COPD patients in their home environment, with and without exacerbation.

DETAILED DESCRIPTION:
In total 130 COPD patients will be included prospectively in this multicenter trial during an inpatient pulmonary rehabilitation program at the Schoen Klinik Berchtesgadener Land, Schönau am Koenigssee, (Germany) or during a stay (inpatient or outpatient) at the Klinikum Nuremberg (Germany).

In general, the study is divided into two parts - study part I, within the duration of the pulmonary rehabilitation program/ hospital stay and study part II, in the home environment (24 weeks).

Study part I:

Visit 1 (day 0, in the clinic) + Visit 2* (day 14+/-5, in the clinic/outpatient)

Each study participant is given a smartphone. Under the guidance of study personnel, data collection of the following parameters is carried out via KAIA mCST App):

* four standardized questions regarding coughing frequency, expectoration, chest tightness and shortness of breath during exercise
* Dyspnea at rest
* Breath sounds via microphone
* Inspiration/expiration length via microphone
* Respiratory rate via smartphone measurements
* Physical performance via the sit-to-stand test (1min) with counting the repetitions and checking the correct execution via smartphone camera
* Gait analysis (2x 10 steps walking) via acceleration sensors of the smartphone or via motion tracking by camera during defined gait measurements.

The mCST app takes about 15 minutes to complete.

Additionally, clinical routine data will be collected:

* medical history
* body plethysmography & blood gases
* EKG
* health related quality of life
* dyspnea
* 6-minute walk distance
* 1-minute-sit to stand test

Study part II:

Visits 3 to 26 (week 3 to 26, in participants home environment) From study visit 3 on, participants are observed weekly in their home environment for a total of 24 weeks. No further clinic visits take place. Disease activity is measured weekly as patient reported outcomes using the mCST app (for details see description of visit 1/2, part 1). In addition to the weekly mCST app, patients are invited to fill out daily a symptom diary before going to bed. The symptom diary contains the EXACT questionnaire and an activity questionnaire.

*Visit 2 is optional

ELIGIBILITY:
Inclusion Criteria:

* hospitalisation at Schoen Klinik Berchtesgadener Land or Klinikum Nuremberg
* Chronic obstructive pulmonary disease GOLD A-D
* sufficient german language and samrtphone skills to understand the mCST app
* sufficient good WLAN Connection in the domestic environment

Exclusion Criteria:

* presence of comorbidities which could interfere the course of the trial (e.g. cognitive deficits, neurological or orthopedic diseases)
* significant mental illness, legal incapacity or limited legal capacity
* patients who are unable or unwilling to perform the study activities acording to the protocol

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation between usual physical exercise tests and exercise test measured via mobile COPD status test app (mCST) | Visit 1 (Day 0)
  Correlation between the 6-minute walk test distance (clinical routine) and the number of repetitions of the 1-minute sit-to-stand-test (mCST app)
Correlation between usual physical exercise tests and exercise test measured via mobile COPD status test app (mCST) | if applicable Visit 2 (Day 14)
  Correlation between the 6-minute walk test distance (clinical routine) and the number of repetitions of the 1-minute sit-to-stand-test (mCST app)

SECONDARY OUTCOMES:
Correlation between COPD Assessment test and perception of disease activity measured via mobile COPD status test app (mCST) | weekly up to 26 weeks (Visit 1 to Visit 26)
  Correlation between standardized questions about COPD activity/ symptoms via the mCST app and the COPD Assessment Test
Correlation between modified medical research scale (mMRc) and perception of dyspnea measured via mobile COPD status test app (mCST) | Visit 1 (Day 0)
  Correlation between standardized questions about dyspnea collected via the mCST app and the modified medical research scale
Correlation between modified medical research scale (mMRc) and perception of dyspnea measured via mobile COPD status test app (mCST) | if applicable Visit 2 (Day 14)
  Correlation between standardized questions about dyspnea collected via the mCST app and the modified medical research scale
Correlation between lung function parameters and inspiratory-/expiratory duration measured via mobile COPD status test app (mCST) | Visit 1 (Day 0)
  Correlation between inspiratory-/ expiratory duration via the mCST app and FEV1, RV, TLC, VC
Correlation between lung function parameters and inspiratory-/expiratory duration measured via mobile COPD status test app (mCST) | if applicable Visit 2 (Day 14)
  Correlation between inspiratory-/ expiratory duration via the mCST app and FEV1, RV, TLC, VC
Correlation between mCST app and symptom diary (EXACT questionnaire) | weekly up to 26 weeks (Visit 1 to Visit 26)
  Correlation between standardized questions about COPD activity/symptoms via the mCST app and the EXACT questionnaire, which consists of 14 questions to quantify exacerbations.
Correlation between mCST app and symptom diary (Freiburger activity questionnaire) | weekly up to 26 weeks (Visit 1 to Visit 26)
  Correlation between standardized questions about COPD activity/ symptoms via the mCST app and the Freiburger activity questionnaire, which consists of 12 items and measures the duration and frequency of various basic, everyday and sports activities of the past week
Differences in outcomes of the mobile COPD status test app (mCST) between patients without and with exacerbations during the study period | weekly up to 26 weeks (Visit 1 to Visit 26)
  Change in the mCST app parameters during the trial period in stable COPD patients an COPD patients with an acute exacerbations during the study period

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Klinikum Nürnberg, Klinik für Innere Medizin3, Schwerpunkt Pneumologie, Nuremberg
  - Klinikum Berchtesgadener Land, Schön Kliniken, Schönau am Königssee

IPD SHARING:
Plan to Share IPD: No